CLINICAL TRIAL: NCT05404178
Title: Turkish Validity-Reliability Study of the Diabetic Foot Self-Care Questionnaire
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, İbrahim Caner Di̇ki̇ci̇, Lecturer, Harran University
Other Study IDs: 25746723
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Diabete Type 2; Diabetic Foot
Keywords: Diabete Type 2; Diabetic Foot; Validity and reliability
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Type 2 diabetes group — This is a single-center, prospective, observational study. The assessment and reporting will be followed the Consensus-Based Standards for the Selection of Health Status Measurement Instruments (COSMIN) checklist.
  Other Names: Assesment

SUMMARY:
The aim of this study is to evaluate the translation, cross-cultural adaptation and psychometric properties of the Diabetic Foot Self-Care Questionnaire in patients with primary Type 2 Diabetes.

DETAILED DESCRIPTION:
This study will be conducted in descriptive type. The population of the research will be patients with diabetic foot in the Endocrinology clinic and polyclinic of the University Hospital. The sample of the study will consist of patients who meet the research criteria and agree to participate in the research. The data collection tools of the study are the patient questionnaire (19 questions), the Diabetic Foot Self-Care Questionnaire (16 questions) and the Foot Care Behavior Scale, by scanning the literature by the researchers.

English Turkish translations will be made before starting the research. Afterwards, expert opinion will be taken for the suitability of the scale items. Then, the Turkish scale items will be translated back into English and the linguist's opinion will be taken that the scale can be applied. Language and content validity will be done for the scale form. The scale items will be translated into Turkish and expert opinions will be taken. Then, the Turkish scale items will be translated back into English and the linguist's opinion will be taken that the scale can be applied. Language validity and content validity will be done in the study. Explanatory Factor Analysis will be applied for the validity of the questionnaire. Kaiser Meyer Olkin(KMO) Test, which measures the adequacy of sample size as antecedent tests, and Bartlett's Test For Sphericity will be used to test sphericity. Factor Analysis Principal Component Analysis Method will be applied.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years old
* Having Type 2 Diabetes and having a diabetic foot ulcer.
* Volunteering to participate in the research.

Exclusion Criteria:

* Have a communication problem
* Presence of lower extremity amputation
* Presence of any ulcer other than diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Diabetic Foot Self-Care Questionnaire | Baseline
  The Turkish validity and reliability of a scale consisting of 16 questions created to evaluate self-care in patients with diabetic foot has not been determined. The survey is divided into 3 areas. Areas 1 to 6 are self-care areas, Items 7 to 11 are self-management areas, and areas 12 to 16 are self-exploration areas.

SECONDARY OUTCOMES:
Foot Care Behavior Scale | Baseline
  It was created to develop foot self-care behaviors in diabetes. The scale, which is a 5-point Likert type scale, is scored according to agree-disagreement (1= Never, 2= Sometimes, 3= Sometimes, 4= Often, and 5= Always) and consists of 15 items. The lowest score that can be obtained from the scale, which evaluates foot care behavior as a single dimension, is 15 and the highest score is 75. An increase in the scale score indicates that the individual's foot self-care behaviors are better.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim C Di̇ki̇ci̇, MSc, Study Director — Harran University; Zeynal Yasacı, MSc, Study Chair — Harran University; Derya Tülüce, PhD, Study Chair — Osmaniye Korkut Ata University
Locations (1):
- Harran University, Sanliurfa, Türki̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No